CLINICAL TRIAL: NCT00985101
Title: Study of the Significance of Mitochondrial Dysfunction for Development of Diabetic Complications
Brief Title: Study of Cellular Impairments Involved in Diabetic Complications
Acronym: diabmito I
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Naestved Hospital (Other)
Responsible Party: Chief Physician, M.D., DMSc. Ass. prof. Jan Kvetny, Department of Internal Medicine & Faculty of Health Sciences, University of Copenhagen
Other Study IDs: SJ-109
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- diabetes no complications
- diabetes with complications

SUMMARY:
The purpose of this study is to examine if an early detectable dysfunction in a cellular component (mitochondria) may predict complications in diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus

Exclusion Criteria:

* Age below 18 yrs
* Psychiatric disease
* Other metabolic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient diabetes clinic Naestved Hospital, denmark
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-04

PRIMARY OUTCOMES:
endothelial damage | 3 times pr years